CLINICAL TRIAL: NCT02753933
Title: An Observational Study to Evaluate Referral From General Practitioners (GPs) to: 1) Direct Access to Magnetic Resonance Imaging (MRI); and 2) the Neurology Department for the Management of Patients With Chronic Headache.
Brief Title: Direct Access to MRI and Neurology Referrals for the Management of Patients With Chronic Headache.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: MRI headache v2.0
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Chronic Headache
MeSH Terms: conditions — Headache Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MRI scan: Direct referral from Primary Care (GPs) to an MRI scan as the initial Secondary Care point of contact.
  Interventions: Other: MRI scan
- Neurology Appointment: Referral from Primary Care (GPs) to Neurology Services in Secondary Care as the initial Secondary Care point of contact.
  Interventions: Other: Neurology Appointment

INTERVENTIONS:
Other: MRI scan — MRI head scan to be performed as the first Secondary Care contact.
  Groups: MRI scan
Other: Neurology Appointment — Outpatient appointment with Neurologist as the first Secondary Care contact
  Groups: Neurology Appointment

SUMMARY:
This study aims to evaluate whether direct access from General Practitioners (GPs) to Magnetic Resonance Imaging (MRI) for patients with chronic headache decreases overall NHS costs and increases patient satisfaction compared to clinical practice with referral to Neurology Services.

DETAILED DESCRIPTION:
Headache is the most common symptom reported in the community, affecting more than 90% of the population at some point in their lifetime. Despite the low level of referrals to secondary care (as most patients tend to be managed within primary care), the absolute number of headache episodes (due to its high prevalence) makes headache the most frequently listed reason for referral to the Neurologist and thus, utilises precious capacity that is severely constrained.

In order to support future management of this chronic condition, this study aims to evaluate existing clinical pathways in the management of patients with chronic headache - either referral to the Neurology Department or direct access to Imaging. Participants will be followed-up for a period of 12 months after the initial Secondary Care episode (either an MRI scan or Neurology appointment). Costs from the NHS perspective and self-perceived patient quality of life will be assessed and cost per patient and cost-effectiveness analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Every patient aged 16 years or over with: i) chronic headache as a primary cause that has lasted ≥ 15 days per month for more than 3 months; and ii) referred from GP practices to GSTT, either directly referred to an MRI exam or a Neurology outpatient appointment.

Exclusion Criteria:

* Children under the age of 16;
* Patients with red flags as defined in NICE guideline CG150;
* Patients without chronic primary headache, i.e. a headache that has not persisted for ≥ 15 days per month for more than 3 months
* Patients with headache referred through the two week wait list;
* Patients who lack capacity to give consent or participate in the study;
* Patients not fluent in English;
* Prisoners;
* Patients that are already taking part in a clinical trial of an investigational medicinal products (CTIMPs).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic headache referred from Primary Care to Secondary Care to either an MRI scan or a Neurology outpatient appointment.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
6-month cost analysis per patient referred to either MRI or Neurology (measured in £ per patient) | 6 months after the initial episode at Secondary Care (either an MRI scan or Neurology Outpatient appointment)
  The primary objective is to evaluate whether direct access from General Practitioners (GPs) to Magnetic Resonance Imaging (MRI) for patients with chronic headache is associated with cost-savings at 6 months after the initial episode at Secondary Care (either an MRI scan or a Neurology Outpatient appointment) compared to clinical practice with referral to the Neurology Department.

SECONDARY OUTCOMES:
12-month cost analysis per patient referred to either MRI or Neurology (measured in £ per patient) | 12 months after the initial episode at Secondary Care (either an MRI scan or Neurology Outpatient appointment)
  This secondary objective is aimed at evaluating whether direct access from General Practitioners (GPs) to Magnetic Resonance Imaging (MRI) for patients with chronic headache is associated with cost-savings at 12 months after the initial episode at Secondary Care (either an MRI scan or a Neurology Outpatient appointment) compared to clinical practice with referral to the Neurology Department.
6-month cost-effectiveness analysis per patient referred to either MRI or Neurology (measured in £ per QALY) | 6 months after the initial episode at Secondary Care (either an MRI scan or Neurology Outpatient appointment)
  This secondary objective is aimed at evaluating whether direct access from General Practitioners (GPs) to Magnetic Resonance Imaging (MRI) for patients with chronic headache is cost-effective at 6 months after the initial episode at Secondary Care (either an MRI scan or a Neurology Outpatient appointment) compared to clinical practice with referral to the Neurology Department.
12-month cost-effectiveness analysis per patient referred to either MRI or Neurology (measured in £ per QALY) | 12 months after the initial episode at Secondary Care (either an MRI scan or Neurology Outpatient appointment)
  This secondary objective is aimed at evaluating whether direct access from General Practitioners (GPs) to Magnetic Resonance Imaging (MRI) for patients with chronic headache is cost-effective at 12 months after the initial episode at Secondary Care (either an MRI scan or a Neurology Outpatient appointment) compared to clinical practice with referral to the Neurology Department.
Patient satisfaction associated with both clinical pathways (direct referral to MRI or Neurology) | 6 months
  To evaluate and compare the levels of patient satisfaction associated with the two pathways: i) with direct access to MRI from Primary Care; and ii) with referral to the Neurology Department. A patient satisfaction questionnaire will be used to quantify patient satisfaction at 6 months.
Patient's self perceived quality of life - measured using EQ-5D-5L questionnaire | 6 months
  This objective aims to evaluate the patient's self-perceived quality of life associated with both pathways using a standard questionnaire (EQ-5D-5L).
Patient's self perceived quality of life - measured using HIT-6 questionnaire | 6 months
  This objective aims to evaluate the patient's self-perceived quality of life associated with both pathways using a standard headache-specific questionnaire (HIT-6 questionnaire).
Patient's self perceived quality of life - measured using MIDAS questionnaire | 6 months
  This objective aims to evaluate the patient's self-perceived quality of life associated with both pathways using a standard headache-specific questionnaire (MIDAS questionnaire).
Time-off work (measured in half days) due to chronic headache | 12 months
  To evaluate the headache burden and time-off work (both measured in half days) due to the chronic headache associated with the pathway with direct access to MRI compared with referral to the Neurology Department.

CONTACTS AND LOCATIONS:
Overall Officials: Asif Mazumder, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rua T, Mazumder A, Akande Y, Margariti C, Ochulor J, Turville J, Razavi R, Peacock JL, McCrone P, Goh V, Shearer J, Afridi S. Management of chronic headache with referral from primary care to direct access to MRI compared with Neurology services: an observational prospective study in London. BMJ Open. 2020 Oct 16;10(10):e036097. doi: 10.1136/bmjopen-2019-036097. PMID 33067273